CLINICAL TRIAL: NCT01033760
Title: Optimisation of Primary HIV1 Infection Treatment (ANRS 147 OPTIPRIM)
Brief Title: Optimisation of Primary HIV1 Infection Treatment(ANRS 147 OPTIPRIM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-014742-28; EudraCT (Registry Identifier: 2009-014742-28)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: HIV-1 Infections
Keywords: Primary HIV-1 infection; antiretroviral treatment; HIV reservoirs; HIV-DNA levels; randomized; Treatment Naive
MeSH Terms: interventions — Raltegravir Potassium; Maraviroc; Darunavir; Ritonavir; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm 1 (Experimental): darunavir, ritonavir, emtricitabine/tenofovir, maraviroc, raltegravir
  Interventions: Drug: raltegravir; maraviroc; darunavir; ritonavir; tenofovir/emtricitabine
- arm 2 (Active Comparator): darunavir, ritonavir, emtricitabine/tenofovir
  Interventions: Drug: darunavir; ritonavir; emtricitabine/tenofovir

INTERVENTIONS:
Drug: raltegravir; maraviroc; darunavir; ritonavir; tenofovir/emtricitabine — raltegravir (Isentress®): 400 mg bid. maraviroc (Celsentri®): 150 mg bid. darunavir (Prezista®): 800 mg QD. ritonavir tablet (Norvir®): 100 mg QD. tenofovir/emtricitabine (Truvada®): one 245/200 mg tablet QD.
  Arms: arm 1
Drug: darunavir; ritonavir; emtricitabine/tenofovir — darunavir (Prezista®): 800 mg QD. ritonavir tablet (Norvir®): 100 mg QD. tenofovir/emtricitabine (Truvada®): one 245/200 mg tablet QD.
  Arms: arm 2

SUMMARY:
The purpose of this trial is to assess the impact of raltegravir, maraviroc, darunavir/r, and Truvada® (emtricitabine/tenofovir) vs. darunavir/r and Truvada® on cell-associated HIV-DNA levels in patients with primary HIV-1 infection.

DETAILED DESCRIPTION:
Primary HIV-1 infection is characterized by a phase of intense replication, with a quick dissemination and early changes in the immune system. During primary HIV-1 infection, damages to MALT and GALT promotes a chronic cell activation, which participates in a progressive decay of immune functions.

After HAART initiation, the magnitude and rapidity of cell-associated HIV-DNA decrease are significantly higher in patients with primary HIV-1 infection than in patients with chronic infection (Ngo Giang Huong, AIDS 2004).

We hypothesize that an early intervention at different levels of viral replication with potent and well-tolerated new drugs may have a greater impact on cell-associated HIV-DNA levels than conventional triple-drug HAART.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute or primary HIV-1 infection
* Acute infection: negative or slightly positive Elisa, with negative or incomplete western-blot (0 or 1 antibody) and positive HIV-RNA and/or positive Ag p24.
* Primary infection: positive Elisa with incomplete Western-blot (≥ 2 and < 5 antibodies with the presence of anti-p24 antibodies associated with an anti-gp160 or an anti-gp120 or an anti-gp41antibody) and positive HIV-RNA.
* Symptomatic Primary infection or CD4 <500/mm3
* written informed consent
* ≥ 18 years old

Exclusion Criteria:

* Prior post exposure antiretroviral treatment within six months before enrolment
* Pregnancy or breast-feeding
* HIV-2 infection
* Current malignancy
* Prothrombin time < 50%
* Creatinine clearance < 60 ml/min
* ASAT, ALAT or bilirubin ≥10*N
* Platelets < 25000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-04; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To compare the 24-month impact of maximized vs. conventional HAART- on HIV reservoirs, as assessed by cell-associated HIV-DNA levels, in patients with acute or primary HIV-1 infection | 24 months

SECONDARY OUTCOMES:
Plasma HIV-RNA levels and proportion of patients with plasma viral load < 50 copies/ml at M12, M24 and M30 | 30 months
Plasma HIV-RNA levels and proportion of patients with plasma viral load < 5 copies/ml at M24 | 24 months
Changes in cell-associated HIV-DNA between baseline and M24 | 24 Months
Evolution of the CD4 and CD8 between D0 and M24 | 24 months
Tolerability of trial treatments | 24 months
Number and type of ARV mutations in virological failures and change in CCR5 tropism | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CHERET, PH, Principal Investigator — Tourcoing Hospital; Caroline LASCOUX-COMBE, PH, Principal Investigator — Saint Louis Hospital, Paris; Laurence MEYER, Professor, Study Chair — Methodologist, INSERM U1018; Bruno HOEN, Professor, Principal Investigator — Saint Jacques Hospital, CHU Besançon; Isabelle RAVAUX, PH, Principal Investigator — Conception Hospital, Marseille; Christine ROUZIOUX, Professor, Principal Investigator — Virology Investigator, Necker Hospital Paris; Alain VENET, PH, Principal Investigator — Immunology Investigator, INSERM U1012 Bicêtre; Daniel OLIVE, Professor, Principal Investigator — Immunology Investigator, Cancerology Institut Marseille; Gianfranco PANCINO, PH, Principal Investigator — Immunology Investigator, Pasteur Institut Paris; Brigitte AUTRAN, Professor, Principal Investigator — Immunology Investiigator, INSERM U543 Paris
Locations (1):
- Hôpital Gustave Dron, Tourcoing, France

REFERENCES:
- [Derived] Cheret A, Durier C, Melard A, Ploquin M, Heitzmann J, Lecuroux C, Avettand-Fenoel V, David L, Pialoux G, Chennebault JM, Muller-Trutwin M, Goujard C, Rouzioux C, Meyer L; ANRS OPTIPRIM study group. Impact of early cART on HIV blood and semen compartments at the time of primary infection. PLoS One. 2017 Jul 14;12(7):e0180191. doi: 10.1371/journal.pone.0180191. eCollection 2017. PMID 28708873
- [Derived] Cheret A, Nembot G, Melard A, Lascoux C, Slama L, Miailhes P, Yeni P, Abel S, Avettand-Fenoel V, Venet A, Chaix ML, Molina JM, Katlama C, Goujard C, Tamalet C, Raffi F, Lafeuillade A, Reynes J, Ravaux I, Hoen B, Delfraissy JF, Meyer L, Rouzioux C; OPTIPRIM ANRS Study Group. Intensive five-drug antiretroviral therapy regimen versus standard triple-drug therapy during primary HIV-1 infection (OPTIPRIM-ANRS 147): a randomised, open-label, phase 3 trial. Lancet Infect Dis. 2015 Apr;15(4):387-96. doi: 10.1016/S1473-3099(15)70021-6. Epub 2015 Feb 18. PMID 25701561